CLINICAL TRIAL: NCT05523830
Title: Estimation of Energy Expenditure and Physical Activity Classification With Wearables
Acronym: EEPAC
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Ministry of Economic Affairs (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL80580.068.22
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Energy Metabolism; Algorithms
Keywords: Energy expenditure; Physical Activity; Wearables
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Urine samples for deutrium dilution analysis to asses total body water
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Subjects: 56 healhty subjects will be recruited for the current study
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
Regular physical activity (PA) is proven to help prevent and treat several non-communicable diseases such as heart disease, stroke, and diabetes. Intensity is a key characteristic of PA that can be assessed by estimating energy expenditure (EE). However, the accuracy of the estimation of EE based on accelerometers are lacking. It has been suggested that the addition of physiological signals can improve the estimation. How much each signal can add to the explained variation and how they can improve the estimation is still unclear.

The goal of the current study is twofold:

to explore the contribution of heart rate (HR), breathing rate (BR) and skin temperature to the estimation of EE develop and validate a statistical model to estimate EE in simulated free-living conditions based on the relevant physiological signals.

DETAILED DESCRIPTION:
Physical activity (PA) is defined as any bodily movement produced by skeletal muscle that requires energy expenditure. The scientific evidence for the beneficial effects are irrefutable. Regular PA is proven to help prevent and treat several non-communicable diseases such as heart disease, stroke, diabetes and different forms of cancer.

PA is a complex behaviour that is characterized by frequency, intensity, time and type (FITT). In order to understand the effect of PA on health and our general well-being, it is essential to monitor all four characteristics of PA. A PA classification algorithm can assess the amount of time spent in different body postures and activity. Making it possible to assess frequency, time and type. In order to completely characterize PA, intensity needs to be estimated. This can be done by the estimation of energy expenditure (EE).

Wearables play a crucial role in the monitoring of PA. They are practical way to collect objective PA data in daily life, in an unobtrusive way, at a relatively low cost. Furthermore they can be applied as a motivational tool to increase PA. Accelerometry has been routinely used to quantify PA and to predict EE using linear and non-linear models. However, the relationship between EE and acceleration differs from one activity to another. For example, cycling can generate the same acceleration amplitude as running, but the EE may differ greatly. It is clear that acceleration alone has a limited accuracy to estimate EE from different activities.

Improving the estimation of EE could be achieved by first classifying the activity type. For each type of activity, different estimations can be used. There are numerous methods to classify PA and estimate EE. Literature describes the use of regression based equations combined with cut-points, linear models, non-linear models, decision trees, artificial neural networks, etc. It is still unclear what would be the best method to estimate EE, not to mention which features would contribute to the model.

Another possibility is to add a relevant bio-signal to the estimation model. Heart rate, breathing rate, temperature are all signals that have a response related to an increase in PA. Heart rate has been used previously to improve the EE estimation in combination with accelerometry. The breathing rate and temperature could contribute to the estimation of EE is still unclear.

Therefore, the goal of the current study is twofold. Firstly, to explore the contribution of different variables (physiological signals) to the estimation of EE and the classification of PA. Secondly, develop and validate a model to estimate EE and classify PA in simulated free-living conditions based on the relevant variables.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 64 years
* Provided written informed consent
* Able to be physically active assed with PAR-Q+

Exclusion Criteria:

* A contraindication to physical activity
* A contraindication to wearing wearables, fixed by a hypoallergenic plaster
* Chronic disease
* A pace maker or any chest-implanted device

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults that are able to be physically active
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure Estimation Model | 1.5 years
  The primary objective of this study is to develop and validate an energy expenditure estimation and physical activity classification algorithm based on wearable sensors. To do so the relevant signals contributing to the classification of physical activity and the estimation of energy expenditure will be identified.

SECONDARY OUTCOMES:
Heart rate (variability) algorithm | 1.5 years
  Design and validate a heart rate (variability) algorithm
  - Investigate the feasibility of modelling the instantaneous energy expenditure
Contribution of different bio signals to the estimation of energy expenditure | 1.5 years
  Assess the contribution of different bio signals to the estimation of energy expenditure
Instantaneous energy expenditure | 1.5 years
  Investigate the feasibility of modelling the instantaneous energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Guy Plasqui, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD is undecided